CLINICAL TRIAL: NCT06485011
Title: Comparison Of Outcome Of Wound Closure After Thyroid Surgery With And Without Platysma Suturing
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children Hospital and Institute of Child Health, Lahore (Other)
Responsible Party: Principal Investigator, Muhammad Adeel Ashiq, Principal Investigator, Children Hospital and Institute of Child Health, Lahore
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Adeel7
Record Dates: First submitted 2024-06-26; First posted 2024-07-03 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-06

CONDITIONS: Pain, Acute Postoperative
Keywords: Thyroid surgery; scar; visual analog scale
MeSH Terms: conditions — Pain, Postoperative; Cicatrix

STUDY DESIGN:
Intervention Model Description: 2 groups included
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- With Platysma suturing (Experimental): platysma muscle was sutured in this group
  Interventions: Procedure: Paltysma suturing
- Without Platysma suturing (Experimental): platysma muscle was not sutured in this group
  Interventions: Procedure: Without Platysma suturing

INTERVENTIONS:
Procedure: Paltysma suturing — platysma muscle was sutured in this group with vicryl
  Arms: With Platysma suturing
Procedure: Without Platysma suturing — platysma muscle was not sutured in this group
  Arms: Without Platysma suturing

SUMMARY:
Comparison Of Outcome Of Wound Closure After Thyroid Surgery With And Without Platysma Suturing in terms of wound scar and pain.

DETAILED DESCRIPTION:
This randomized controlled trail was conducted at Surgical Ward from January 2021 to July 2021.

Materials and Methods Total 72 patients (indicated for thyroid surgery) who were fulfilling the inclusion criteria were enrolled. Patients were divided randomly into two groups by using lottery method. In Group A patients wound closure was done without Platysma Suturing and in Group-B patients wound closure was done with Platysma Suturing. Pain assessment was done with the help of VAS after surgery (6, Hours, 24 hours, 48 hours). Scar assessment was carried out with the help of POSAS. All this information was noted by the researcher himself and noted on a well-designed questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* : Both men and women patients in the age range (20-70 years) undergoing primary thyroid surgery were included.

Exclusion Criteria:

* Patients with disorders of wound healing, diabetes mellitus, Pre-operative known malignant condition, history of neck surgery or not willing to participate in the study were excluded.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 72 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2021-07-01 (Actual); Study Completion 2021-09-01 (Actual)

PRIMARY OUTCOMES:
Post operative Pain | 48 hours
  Pain assessed on visual analogue scale. higher the VAS score means more pain and lower score mean less pain

CONTACTS AND LOCATIONS:
Overall Officials: Adeel Ashiq, MS, Principal Investigator — The Children Hospital
Locations (1):
- The Children Hospital, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No
No plan of sharing